CLINICAL TRIAL: NCT05902091
Title: Neurophysiology-based Intervention Program in Sportive Children With Foot Dysfunction
Brief Title: Neurophysiology-based Intervention of Foot Dysfunction in Sportive Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Jitka Marenčáková, Postdoc researcher, Charles University, Czech Republic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UKFTVS_LSM_02
Record Dates: First submitted 2023-05-23; First posted 2023-06-13 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Flatfoot, Flexible; Sports Physical Therapy; Child Development
MeSH Terms: conditions — Flatfoot

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercising participants (Experimental): Participants will receive 4 weeks of neurophysiology-based intervention, forty-five minutes of individual session, twice a week.
  Interventions: Behavioral: Neurophysiology-based intervention

INTERVENTIONS:
Behavioral: Neurophysiology-based intervention

SUMMARY:
The goal of the clinical trial study is to test the effect of the individual complex physiotherapy intervention program in the children actively playing soccer with flatfoot or valgus foot.

The aims are:

1. see if the medial longitudinal arch will by actively more higher after the intervention
2. see if the type of the foot will change toward more neutral type after the intervention
3. see if the transfer of the centre of body mass through the foot during the gait will directed in more neutral line after the intervention

The participants will undergo clinical assessment of short kinesiology assessment visually in underwear and barefoot. Then Participant will be tested for balance test in narrow stance with open and closed eyes, and single.leg stance with open eyes on the pressure mat. Finally, participant will walking in self-selected normal speed through the gait pressure mat. Eaxh procedure will be measured twice, before the program start and after the 4 weeks when the program finish. Researchers will compare these two measurement for the changes.

DETAILED DESCRIPTION:
The aim of the study was to evaluate the effect of the neurophysiology-based (NB) intervention program in sporting children with foot problems. The NB intervention composed from evidence based and neurophysiology-based methods: 1) Janda´s sensorimotor stimulation, 2) Dynamic neuromuscular stabilisation concept (DNS), 3) Toe and foot muscle strengthening, 4) foot support base related exercises, and 5) somatic-sensory facilitation techniques. The proposed NB intervention lasted 4 weeks with each 45minutes long session twice a week. Each session was leaded by experienced physiotherapist in clinical practice gym, in one-to-one regime to ensure quality of the exercising, using progressive steps and some additional balance pads and small ball. The research assessments were conducted pre- and post-intervention (T0 and T4) and consisted of personal data and health questionnaires (name, date of the birth, laterality, shoe size, diseases, injuries and surgery), clinical examining (standing posture, core stabilisation function in supine position, foot posture index), laboratory testing (postural stability and normal walking on pressure mat). Data were edited, analysed and compared pre- and post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* age 9-10 years
* playing football at least for one year and train twice a week
* FPI above 5
* CSI above 45.1%

Exclusion Criteria:

* acute pain, injury
* injury of musculoskeletal system (past 6 months)
* infectious disease
* cardiovascular, metabolic, neurologic or orthopaedic diseases
* active wearing the orthotic devices or aids or barefoot shoes
* previous surgery on the lower limbs or pelvis

Ages: 9 Years to 10 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2016-06-10 (Actual); Primary Completion 2017-09-05 (Actual); Study Completion 2018-09-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline Foot type at 4 weeks | at baseline and in 4 weeks
  The foot type was assessed using the reliable and valid clinical test Foot posture index (6-FPI) which examine 6 items of the foot: talar head position, inversion/eversion of the calcaneus, talonavicular bulging, medial longitudinal arch height, forefoot abd/adduction, each by the point 0 for neutral, +1 and +2 for pronated, and -1 and -2 for supinated position as defined by Redmont et al. (2008). Total score of the 6 items defines foot type as neutral (0 to +5), pronated (+6 to +9), over-pronated (+10 to +12), supinated (-1 to -4) and over-supinated (-5 to -12).
Change from baseline Medial longitudinal arch height at 4 weeks | at baseline and in 4 weeks
  The medial longitudinal arch height (MLAH) was assessed by Chippaux-Smirak index (CSI) from digital foot print obtained from pressure mat during single-leg standing. The software Kinovea was used for the normalization the foot print to real foot size and measuring the widest part of the forefoot and the narrowest part of the midfoot in millimeters. Finally, the index was calculated: the narrowest part was divided by widest part and multiply by 100 to obtain total percentage. Total percentage of the CSI ranges in 5 types of MLAH: high 0-0.1%, normal 0.1-29.9%, transitional 30-39.9%, lowered 40-45%, mild flat 45.1-50%, moderate flat 50.1-60%, severe flat 60.1-100% (Onodera et al., 2008; Nikolaidou and Boudolos, 2006).
Change from baseline Foot dynamic function at 4 weeks | at baseline and in 4 weeks
  The foot dynamic function was measured by Centre of pressure excursion index (CPEI) during normal walking on pressure platform RS Footscan (Gait 7.7). The imposed digital footprint with centre of pressure (COP) trajectory was firstly normalised for the real foot size and measured in software Kinovea to obtain the foot measures: Line A connect the initial point and final point of the COP trajectory, line B was drawn perpendicular to the line A in the widest part of the forefoot, line C was a partial section of the line B between crossing points with line A and COP trajectory. Final calculation of CPEI was done: Line C divided by line B multiplied 100 to obtain total percentage. According to previous studies (Hillstrom et al., 2013; Song et al., 1996), the sample results were divided into thirds: CPEI 10-24.9% for over-pronation, CPEI 25-34.9% for optimal function, and CPEI above 35% for supinated function.
Change from baseline Postural stability at 4 weeks | at baseline and in 4 weeks
  The postural stability function in single-leg stance was measured on pressure platform RS Footscan (Balance 7.6). Participant stood up on the mat 1.5 m far from the wall, watching the point on the wall in the height of his eyes and flexed non-tested leg up to 90° with thigh still in vertical position. Participant was instructed to stand steadily without moving for 60 s with eyes open. After the rest, participant repeated the same measurement on the other side. Centre of pressure path (COPP) length in millimeters was obtained for both legs.
Core stabilization function | at baseline
  The core stabilization function was assessed by clinical test according to protocol of dynamic neuromuscular stabilisation concept (Kolar et al., 2009) in developmental kinesiology position in supine with legs flexed and raised up and experienced physiotherapist observed the quality of the muscle coordination in stabilisation of the trunk and abdominal wall. The quality of the function was defined as these: 1) optimal function (not co-movements of the region, homogenous abdominal wall, harmonic activation aóf all local and global stabilisers), 2) weakened function (not homogenous abdominal wall, light lumbar movement up) and 3) dysfunction with diastasis (insufficiency of the deep abdominal muscle, over-activation m. rectus abdominis, lumbar spine above the ground, movement and instability of the whole region, diastasis).

CONTACTS AND LOCATIONS:
Overall Officials: František Zahálka, prof., Ph.D., Study Director — Faculty of Physical Education and Sport, Charles University; Jitka Marenčáková, Ph.D., Principal Investigator — Faculty of Physical Eduction and Sport, Charles University
Locations (1):
- Faculty of Physical Education and Sport, Charles University, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Yes
It is planned that selected anonymised data will be published in open access research journal and other individual anonymised data just for the request.
Supporting Information: Study Protocol
Time Frame: 1 year from the public registration.
Access Criteria: Researchers can apply for the anonymised dataset by the email to investigator, only for the reasoned request.